CLINICAL TRIAL: NCT06448624
Title: Effect of Single Dose & Intrapocket Prophylactic Antibiotic to Cardiac Implantable Electronic Device-related Infection & Biomarkers
Brief Title: Biomarkers & Infection After Prophylactic Antibiotic in Cardiac Implantable Electronic Device Implantation
Acronym: BI-PACED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Collaborators: Dr. Kariadi General Hospital Medical Center (Other)
Responsible Party: Principal Investigator, Pipin Ardhianto, Principal investigator, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: No.16114/EC/KEPK-RSDK/2024
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Heart Block; CIED Related Infection; CIED-related Infections; Antibiotic Prophylaxis; Biomarkers
Keywords: heart block; CIED related infection; antibiotic prophylaxis; biomarkers
MeSH Terms: conditions — Heart Block | interventions — sultamicillin

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Placebo Comparator): Ampicillin sulbactam 1.5 gram IV preimplantation + ampicillin sulbactam 1.5 gram intrapocket + placebo for 3 days after implantation
  Interventions: Drug: Placebo 3 days
- Control (Experimental): Ampicillin sulbactam 1.5 gram IV preimplantation + ampicillin sulbactam 1.5 gram intrapocket + ampicillin sulbactam 1.5 gram IV BID for 3 days after implantation
  Interventions: Drug: Ampicillin sulbactam 3 days

INTERVENTIONS:
Drug: Ampicillin sulbactam 3 days — Ampicillin sulbactam 1.5 gram IV BID for 3 days after CIED implantation
  Arms: Control
Drug: Placebo 3 days — Placebo for 3 days after CIED implantation
  Arms: Intervention

SUMMARY:
Effect of single dose & intrapocket prophylactic antibiotic to cardiac implantable electronic device-related infection & biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Indication of CIED implantation
* No infection at the time of implantation

Exclusion Criteria:

* Refuse to participate in the study
* Allergy to ampicillin sulbactam
* CIED debridement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of CIED-related infection | Baseline, 3 days, 7 days, and 28 days
  Incidence of superficial infection, pocket infection, infective endocarditis, or rehospitalization

SECONDARY OUTCOMES:
Level of Presepsin | Baseline and 24 hours after CIED implantation
  Delta level of Presepsin
Level of Interleukin-6 | Baseline and 24 hours after CIED implantation
  Delta level of Interleukin-6
Level of Procalcitonin | Baseline and 24 hours after CIED implantation
  Delta level of Procalcitonin

CONTACTS AND LOCATIONS:
Locations (1):
- Kariadi Central General Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Waiting for agreement